CLINICAL TRIAL: NCT01227564
Title: A Phase 2, Multicenter, 24-month, Randomized, Third-party Unblinded, Placebo-controlled, Parallel-group Amyloid Imaging Positron Emission Tomography (Pet) And Safety Trial Of Acc-001 And Qs-21 Adjuvant In Subjects With Early Alzheimer's Disease.
Brief Title: Amyloid Imaging And Safety Study Of ACC-001 In Subjects With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2571010; B2571010; 3134K1-2208 (Other: Alias Study Number)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Early Alzheimer's disease; active immunization; amyloid imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar; saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACC-001 3 μg/ QS-21 50 μg (Experimental)
  Interventions: Biological: ACC-001 3 μg/ QS-21 50 μg
- ACC-001 10 μg/ QS-21 50 μg (Experimental)
  Interventions: Biological: ACC-001 10 μg/ QS-21 50 μg
- Placebo- Phosphate buffered saline (PBS) (Placebo Comparator)
  Interventions: Other: Placebo- Phosphate buffered saline (PBS)

INTERVENTIONS:
Biological: ACC-001 3 μg/ QS-21 50 μg — ACC-001 3 μg/ QS-21 50 μg IM on day 1, month 1, month 3, month 6, month 12, and month 18
  Other Names: Vanutide Cridificar
  Arms: ACC-001 3 μg/ QS-21 50 μg
Biological: ACC-001 10 μg/ QS-21 50 μg — ACC-001 10 μg/ QS-21 50 μg IM on day 1, month 1, month 3, month 6, month 12, and month 18
  Other Names: Vanutide Cridificar
  Arms: ACC-001 10 μg/ QS-21 50 μg
Other: Placebo- Phosphate buffered saline (PBS) — Phosphate buffered saline IM on day 1, month 1, month 3, month 6, month 12, and month 18
  Arms: Placebo- Phosphate buffered saline (PBS)

SUMMARY:
This study in individuals with early Alzheimer's disease is designed to assess:(1) safety and tolerability (2) the capacity of ACC-001 and QS-21 adjuvant to reduce brain amyloid load as measured by positron emission tomography (PET) scans.

ELIGIBILITY:
Inclusion Criteria:

* Concern about a change in cognition expressed by the subject or by an informant that knows the subject well
* Mini-Mental State Examination (MMSE) score ≥ 25
* Global Clinical Dementia Rating = 0.5.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's dementia cannot not be made by the site physician at the time of screening.
* Amyloid burden detected on screening brain PET scan.
* Other inclusion criteria apply.

Exclusion Criteria:

* Significant neurological disease other than early Alzheimer's disease
* Major psychiatric disorder or symptom
* Contraindication to undergo brain MRI
* Unstable medical conditions
* Other exclusion criteria apply

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (40):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Banner Boswell Medical Center, Sun City, Arizona
  - Banner Lakes Imaging Center, Sun City, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Southwest PET Institute, Tucson, Arizona
  - University of Arizona, Health Sciences Center - Department of Neurology, Tucson, Arizona
  - Universal Medical Center, Tucson, Arizona
  - Northwest NeuroSpecialists, LLC, Tucson, Arizona
  - Radiology Limited, Tucson, Arizona
  - Pacific Neuroscience Medical Group, Oxnard, California
  - GCRC (Drug administered), New Haven, Connecticut
  - Yale University School of Medicine, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Investigational Drug Service, New Haven, Connecticut
  - Norman S. Werdiger, MD, New Haven, Connecticut
  - Clinical Research Unit, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Georgetown University Medical Center Department of Neurology, Washington D.C., District of Columbia
  - Meridien Research, Brooksville, Florida
  - Florida Neurology Group PL, Fort Myers, Florida
  - Internal Medicine Associates of Lee County, MD, PA, Fort Myers, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Florida Radiology Leasing, Limited Liability Corporation, Fort Myers, Florida
  - Radiology Regional Center, Fort Myers, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Premiere Research Institute (Palm Beach Neurology), West Palm Beach, Florida
  - Massachusetts General Hospital (For PET only), Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Steinberg Diagnostic Imaging, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memory Enhancement Center of America, Incorporated, Eatontown, New Jersey
  - Satatoga PET Associates, Clifton Park, New York
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Baylor College of Medicine, Department of Neurology, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - The Pharmacy Inc., Bennington, Vermont

REFERENCES:
- [Derived] van Dyck CH, Sadowsky C, Le Prince Leterme G, Booth K, Peng Y, Marek K, Ketter N, Liu E, Wyman BT, Jackson N, Slomkowski M, Ryan JM. Vanutide Cridificar (ACC-001) and QS-21 Adjuvant in Individuals with Early Alzheimer's Disease: Amyloid Imaging Positron Emission Tomography and Safety Results from a Phase 2 Study. J Prev Alzheimers Dis. 2016;3(2):75-84. doi: 10.14283/jpad.2016.91. PMID 29210443
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2571010&StudyName=Amyloid%20Imaging%20And%20Safety%20Study%20Of%20ACC-001%20In%20Subjects%20With%20Early%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty study centers in the United States of America participated. One of these did not enroll any participants.
Pre-assignment Details: Participants, who were found eligible, were randomized to 1 of 3 groups in a 1:1:1 ratio between ACC-001 3 μg+QS-21, or ACC-001 10 μg+QS-21, or placebo (which was administrated as phosphate buffered saline [PBS]). The study randomization was stratified based on apolipoprotein E (Apo E) genotype (E4 carrier or non-carrier).
Groups:
- ACC 3 μg+QS-21: Participants received 3 μg of ACC-001 and 50 μg of QS-21. Investigational product was administered by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, 12, and 18 months.
- ACC 10 μg+QS-21: Participants received 10 μg of ACC-001 and 50 μg of QS-21. Investigational product was administered by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, 12, and 18 months.
- Placebo: Participants received PBS. Investigational product was administered by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, 12, and 18 months.
Period: Overall Study
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Started | 22 | 20 | 21
Treated | 22 | 20 | 21
Completed Treatment | 21 (1 participant discontinued treatment due to an adverse event (AE).) | 18 (2 participants discontinued treatment due to no longer willing to participate in study.) | 17 (1 participant stopped treatment due to lack of efficacy, 3 due to no longer willing to participate.)
Completed | 18 (Completed study) | 18 (Completed study) | 15 (Completed study)
Not Completed | 4 | 2 | 6
Not completed — No Longer Willing to Participate | 4 | 2 | 5
Not completed — Participant moved to another town | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 21 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.31) | 68.5 (7.02) | 69.6 (6.82) | 68.3 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 9 | 33
  Male | 11 | 7 | 12 | 30
MMSE Score [Mean (Standard Deviation); unit: score] — The MMSE is a brief, structured examination of cognitive function consisting of the 11 item: Orientation-What, Orientation-Where, Registration-Objects, Attention and Calculation, Recall, Language-Naming, Language-Repetition, Language-Comprehension, Language-Reading, Language-Writing, and Language- Drawing. MMSE total score was the sum of the 11 item scores and it ranges from 0 to 30 with higher score indicating greater cognitive functioning. If any individual item is missing, then the MMSE total score is set to missing.
  score | 27.3 (1.64) | 27.7 (1.63) | 28.0 (1.47) | 27.6 (1.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brain Fibrillar Beta-Amyloid Protein (Aβ) at Week 104 as Measured by Standard Uptake Value Ratios (SUVRs) Over the Composite Regions of Interest (ROIs)
Description: Fibrillar brain Aβ was measured by retention of florbetapir F18 as measured by positron emission tomography (PET) scans. A positive change indicating an improvement from baseline.
Time Frame: 104 weeks
Population: The full analysis set (FAS) population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- Overall ACC + QS21: Participants received either 3 μg of ACC-001 and 50 μg of QS-21 or 10 μg of ACC-001 and 50 μg of QS-21. Investigational product was administered by intramuscular injection into the deltoid muscle at 0, 1, 3, 6, 12, and 18 months.
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
ratio
  Week 52 (N: 22, 19, 41, 20) | 0.009 [-0.042 to 0.060] | 0.017 [-0.039 to 0.073] | 0.013 [-0.025 to 0.051] | 0.011 [-0.043 to 0.065]
  Week 78 (N: 21, 18, 39, 16) | -0.011 [-0.084 to 0.062] | -0.022 [-0.101 to 0.057] | -0.017 [-0.071 to 0.038] | -0.014 [-0.096 to 0.068]
  Week 104 (N: 14, 15, 29, 13) | -0.018 [-0.097 to 0.061] | -0.018 [-0.098 to 0.062] | -0.018 [-0.075 to 0.038] | 0.032 [-0.052 to 0.115]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 52; Test type: Superiority or Other; p = 0.9538, Mixed-Effects Model Repeated Measures — Analysis was two-sided and performed at the 0.05 significance level. No multiplicity adjustments due to multiple endpoints or multiple assessments were applied. Nominal p-values were reported in the analysis; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.075 to 0.071]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 10 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 52; Test type: Superiority or Other; p = 0.8787, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.070 to 0.081]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg or ACC 10 µg + QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 52; Test type: Superiority or Other; p = 0.9544, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.062 to 0.066]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 78; Test type: Superiority or Other; p = 0.9550, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.106 to 0.112]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 10 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 78; Test type: Superiority or Other; p = 0.8874, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.121 to 0.105]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg or ACC 10 µg + QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 78; Test type: Superiority or Other; p = 0.9595, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.099 to 0.095]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.3826, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.164 to 0.064]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 10 µg+QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.3912, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.164 to 0.065]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; A mixed-effect model repeated measures was used, with the baseline measure of average SUVRs over ROIs and Apo E4 Status (Carrier or Non-carrier) as covariates, time, treatment, and treatment*time as fixed effects. Estimates of the adjusted mean differences (test-reference) and corresponding 95% confidence intervals were obtained from the model. ACC 3 µg or ACC 10 µg + QS-21 50 µg was the test treatment and placebo was the reference treatment. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.3221, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.050, 95% CI 2-sided [-0.149 to 0.050]

2. Other Pre Specified Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Aβ x-40
Description: For the majority of the participants, the lumbar puncture for the first CSF sample was collected up to 3 days prior to injection of investigational product. For the participants who had a CSF being already drawn at week 80, no CSF sample was drawn at week 104, nor at the Early termination (ET) visit. For those participants who early terminated the study before week 80, CSF was drawn at ET visit.
Time Frame: Week 80 or Week 104
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 18 | 40 | 17
μg/ml | 192.93 [-652.96 to 1038.82] | 726.74 [-252.11 to 1705.58] | 459.83 [-178.24 to 1097.91] | 144.76 [-816.20 to 1105.71]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; Analysis of Covariance (ANCOVA) was used with baseline assessment and ApoE4 status as covariates, in addition to treatment included in the ANCOVA model; Test type: Superiority or Other; p = 0.9384, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 48.18, 95% CI 2-sided [-1197.07 to 1293.42]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; ANCOVA was used with baseline assessment and ApoE4 status as covariates, in addition to treatment included in the ANCOVA model; Test type: Superiority or Other; p = 0.3945, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 581.98, 95% CI 2-sided [-778.17 to 1942.13]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.5773, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 315.08, 95% CI 2-sided [-812.15 to 1442.30]

3. Other Pre Specified Outcome: Change From Baseline in CSF Aβ x-42
Description: For the majority of the participants, the lumbar puncture for the first CSF sample was collected up to 3 days prior to injection of investigational product. For the participants who had a CSF being already drawn at week 80, no CSF sample was drawn at week 104, nor at ET visit. For those participants who early terminated the study before week 80, CSF was drawn at ET visit.
Time Frame: Week 80 or Week 104
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 18 | 40 | 17
μg/ml | 15.29 [-43.14 to 73.71] | 75.55 [11.89 to 139.21] | 45.42 [1.56 to 89.28] | -8.87 [-75.24 to 57.50]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.5818, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 24.16, 95% CI 2-sided [-63.31 to 111.62]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0648, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 84.42, 95% CI 2-sided [-5.37 to 174.21]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1672, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 54.29, 95% CI 2-sided [-23.47 to 132.05]

4. Other Pre Specified Outcome: Change From Baseline in CSF p-Tau
Description: as for outcome 3
Time Frame: Week 80 or Week 104
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 18 | 40 | 17
μg/ml | -2.32 [-6.80 to 2.15] | -3.47 [-8.43 to 1.49] | -2.90 [-6.14 to 0.35] | 1.03 [-3.89 to 5.96]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3106, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-9.94 to 3.22]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1876, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.51, 95% CI 2-sided [-11.28 to 2.27]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1742, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.93, 95% CI 2-sided [-9.66 to 1.79]

5. Other Pre Specified Outcome: Change From Baseline in CSF Total Tau
Description: as for outcome 3
Time Frame: Week 80 or Week 104
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 18 | 40 | 17
μg/ml | 25.56 [-24.38 to 75.50] | -27.48 [-83.48 to 28.49] | -0.96 [-37.23 to 35.31] | 55.92 [0.97 to 110.86]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4089, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -30.36, 95% CI 2-sided [-103.52 to 42.81]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0327, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -83.40, 95% CI 2-sided [-159.69 to -7.11]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0801, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -56.88, 95% CI 2-sided [-120.82 to 7.06]

6. Other Pre Specified Outcome: Change From Baseline in Plasma Aβ x-40
Description: Site personnel collecting the samples for plasma Aβ (x-40) concentrations and the results were blinded to the participant treatment group assignment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
pg/mL
  Week 12 (N: 22, 19, 41, 20) | 30.42 [-9.80 to 70.63] | 61.70 [18.55 to 104.85] | 46.06 [16.49 to 75.63] | 10.64 [-31.24 to 52.52]
  Week 26 (N: 22, 18, 40, 19) | 150.51 [45.32 to 255.70] | 276.86 [162.50 to 391.66] | 213.68 [135.80 to 291.57] | 51.22 [-61.16 to 163.60]
  Week 52 (N: 22, 18, 40, 19) | 252.87 [166.03 to 339.72] | 313.34 [218.29 to 408.38] | 283.11 [218.68 to 347.53] | 138.74 [45.73 to 231.75]
  Week 78 (N: 22, 17, 39, 17) | 225.15 [105.18 to 345.11] | 344.13 [210.80 to 477.45] | 284.64 [194.93 to 374.35] | 117.31 [-13.47 to 248.08]
  Week 104 (N: 18, 17, 35, 13) | 216.51 [111.67 to 321.35] | 279.00 [164.37 to 393.63] | 247.76 [170.03 to 325.48] | 74.60 [-42.18 to 191.37]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 12; Test type: Superiority or Other; p = 0.4892, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 19.78, 95% CI 2-sided [-37.15 to 76.71]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0915, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 51.06, 95% CI 2-sided [-8.51 to 110.63]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1638, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 35.42, 95% CI 2-sided [-14.88 to 85.72]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 26; Test type: Superiority or Other; p = 0.2006, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 99.29, 95% CI 2-sided [-54.28 to 252.86]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0067, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 225.63, 95% CI 2-sided [65.18 to 386.09]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0204, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 162.46, 95% CI 2-sided [26.05 to 298.87]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 52; Test type: Superiority or Other; p = 0.0766, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 114.13, 95% CI 2-sided [-12.63 to 240.89]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.0181, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 226.82, 95% CI 2-sided [40.23 to 413.41]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.0387, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 167.33, 95% CI 2-sided [9.03 to 325.63]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 78; Test type: Superiority or Other; p = 0.2277, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 107.84, 95% CI 2-sided [-69.29 to 284.97]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0181, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 226.82, 95% CI 2-sided [40.23 to 413.41]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0387, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 167.33, 95% CI 2-sided [9.03 to 325.63]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.0747, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 141.92, 95% CI 2-sided [-14.62 to 298.45]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.0151, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 204.40, 95% CI 2-sided [41.02 to 367.79]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.0161, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 173.16, 95% CI 2-sided [33.25 to 313.07]

7. Other Pre Specified Outcome: Change From Baseline in Volumetric Brain Magnetic Resonance Imaging (MRI) Measurements in Brain Boundary Shift Integral (BBSI)
Description: BBSI measures whole brain atrophy from registered MRI scan pairs, by subtracting the area under the intensity profile across a boundary in the repeat scans from the initial scan (baseline).
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
mL
  Week 10 (N: 22, 20, 42, 20) | -4.100 [-6.850 to -1.351] | -0.952 [-3.840 to 1.935] | -2.526 [-4.544 to -0.509] | -1.449 [-4.316 to 1.419]
  Week 24 (N: 22, 20, 42, 21) | -6.080 [-8.781 to -3.379] | -2.357 [-5.193 to 0.480] | -4.218 [-6.201 to -2.236] | -5.906 [-8.683 to -3.128]
  Week 50 (N: 22, 19, 41, 18) | -12.329 [-15.812 to -8.846] | -5.926 [-9.640 to -2.213] | -9.128 [-11.692 to -6.564] | -10.684 [-14.435 to -6.933]
  Week 76 (N: 21, 17, 38, 15) | -16.579 [-21.361 to -11.797] | -10.802 [-16.022 to -5.582] | -13.690 [-17.242 to -10.138] | -16.196 [-21.573 to -10.818]
  Week 104 (N: 18, 16, 34, 14) | -20.982 [-26.683 to -15.101] | -12.662 [-19.008 to -6.316] | -16.822 [-21.128 to -12.486] | -18.772 [-25.335 to -12.209]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline total brain volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 10; Test type: Superiority or Other; p = 0.1807, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.652, 95% CI 2-sided [-6.570 to 1.267]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8051, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.497, 95% CI 2-sided [-3.515 to 4.508]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5331, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.078, 95% CI 2-sided [-4.519 to 2.364]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline total brain volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p = 0.9274, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-3.990 to 3.641]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.0743, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 3.549, 95% CI 2-sided [-0.360 to 7.458]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.3163, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.687, 95% CI 2-sided [-1.656 to 5.031]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline total brain volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 50; Test type: Superiority or Other; p = 0.5190, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.645, 95% CI 2-sided [-6.721 to 3.430]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.0740, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 4.758, 95% CI 2-sided [-0.476 to 9.991]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.4909, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 5.394, 95% CI 2-sided [-2.937 to 6.049]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline total brain volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 76; Test type: Superiority or Other; p = 0.9151, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.383, 95% CI 2-sided [-7.549 to 6.783]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.1533, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 5.394, 95% CI 2-sided [-2.069 to 12.857]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.4371, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 2.506, 95% CI 2-sided [-3.904 to 8.915]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline total brain volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.6167, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.210, 95% CI 2-sided [-10.999 to 6.579]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p = 0.1844, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 6.110, 95% CI 2-sided [-2.993 to 15.212]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p = 0.6205, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.950, 95% CI 2-sided [-5.888 to 9.878]

8. Other Pre Specified Outcome: Change From Baseline in Volumetric Brain MRI Measurements in Ventricular Boundary Shift Integral (VBSI)
Description: VBSI measures ventricular volume change from registered MRI scan pairs, by subtracting the area under the intensity profile across a boundary in the repeat scans.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
mL
  Week 10 (N: 22, 20, 42, 20) | 0.913 [0.500 to 1.327] | 0.643 [0.209 to 1.076] | 0.778 [0.474 to 1.082] | 0.496 [0.056 to 0.935]
  Week 24 (N: 22, 20, 42, 21) | 1.540 [1.066 to 2.014] | 1.229 [0.732 to 1.726] | 1.385 [1.038 to 1.731] | 1.533 [1.039 to 2.027]
  Week 50 (N: 22, 19, 41, 18) | 3.023 [2.194 to 3.853] | 2.242 [1.364 to 3.120] | 2.632 [2.027 to 3.238] | 3.038 [2.160 to 3.915]
  Week 76 (N: 22, 17, 39, 16) | 4.729 [3.322 to 6.136] | 3.445 [1.923 to 4.967] | 4.087 [3.050 to 5.124] | 4.474 [2.940 to 6.008]
  Week 104 (N: 18, 16, 34, 14) | 6.422 [4.586 to 8.257] | 4.970 [2.999 to 6.941] | 5.696 [4.348 to 7.043] | 5.770 [3.770 to 7.769]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline ventricular volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 10; Test type: Superiority or Other; p = 0.1695, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.418, 95% CI 2-sided [-0.183 to 1.018]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.6331, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.147, 95% CI 2-sided [-0.465 to 0.759]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2907, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.282, 95% CI 2-sided [-0.247 to 0.812]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline ventricular volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p = 0.9846, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.675 to 0.688]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.3845, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.304, 95% CI 2-sided [-1.000 to 0.392]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.6204, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.149, 95% CI 2-sided [-0.748 to 0.450]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline ventricular volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 50; Test type: Superiority or Other; p = 0.9810, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-1.221 to 1.192]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.2034, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.796, 95% CI 2-sided [-2.034 to 0.443]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.4491, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.405, 95% CI 2-sided [-1.469 to 0.659]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline ventricular volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 76; Test type: Superiority or Other; p = 0.8074, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.255, 95% CI 2-sided [-1.827 to 2.337]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p = 0.3444, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.029, 95% CI 2-sided [-3.189 to 1.131]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p = 0.6772, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.387, 95% CI 2-sided [-2.239 to 1.464]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline ventricular volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.6325, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.652, 95% CI 2-sided [-2.063 to 3.367]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.5706, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.800, 95% CI 2-sided [-3.606 to 2.007]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.9513, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.074, 95% CI 2-sided [-2.485 to 2.337]

9. Other Pre Specified Outcome: Change From Baseline in Volumetric Brain MRI Measurements in Hippocampal Boundary Shift Integral (HBSI), Total
Description: Left HBSI and Right HBSI respectively measure the left hippocampal atrophy and the right hippocampal atrophy from registered MRI scan pairs, by subtracting the corresponding area under the intensity profile across a boundary in the repeat scans. HBSI (Total) is defined as the summation of the left HBSI and the right HBSI.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
mL
  Week 10 (N: 22, 20, 42, 20) | -0.056 [-0.097 to -0.015] | -0.016 [-0.059 to 0.027] | -0.036 [-0.066 to -0.006] | -0.041 [-0.084 to 0.002]
  Week 24 (N: 22, 20, 42, 21) | -0.124 [-0.167 to -0.081] | -0.065 [-0.110 to -0.020] | -0.094 [-0.126 to -0.063] | -0.099 [-0.143 to -0.055]
  Week 50 (N: 22, 19, 41, 18) | -0.251 [-0.316 to -0.187] | -0.159 [-0.228 to -0.090] | -0.205 [-0.252 to -0.158] | -0.226 [-0.295 to -0.157]
  Week 76 (N: 22, 17, 39, 16) | -0.357 [-0.460 to -0.253] | -0.255 [-0.368 to -0.142] | -0.306 [-0.383 to -0.229] | -0.334 [-0.448 to -0.219]
  Week 104 (N: 18, 16, 34, 14) | -0.468 [-0.601 to -0.335] | -0.329 [-0.472 to -0.185] | -0.398 [-0.496 to -0.301] | -0.471 [-0.620 to -0.323]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 10; Test type: Superiority or Other; p = 0.6054, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.074 to 0.043]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.4087, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.025, 95% CI 2-sided [-0.035 to 0.084]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.8518, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.046 to 0.056]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p = 0.4216, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.085 to 0.036]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.2730, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.028 to 0.097]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.8549, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.048 to 0.058]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 50; Test type: Superiority or Other; p = 0.5847, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.120 to 0.068]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.1740, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.067, 95% CI 2-sided [-0.030 to 0.163]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.6255, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 0.020, 95% CI 2-sided [-0.063 to 0.103]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 76; Test type: Superiority or Other; p = 0.7658, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.023, 95% CI 2-sided [-0.177 to 0.131]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.3309, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.082 to 0.240]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.6872, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.110 to 0.166]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.9752, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.196 to 0.202]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.1715, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.143, 95% CI 2-sided [-0.064 to 0.349]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.4145, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [-0.105 to 0.250]

10. Other Pre Specified Outcome: Change From Baseline in Volumetric Brain MRI Measurements in HBSI, Left
Description: Left HBSI measures the left hippocampal atrophy from registered MRI scan pairs, by subtracting the corresponding area under the intensity profile across a boundary in the repeat scans.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
mL
  Week 10 (N: 22, 20, 42, 20) | -0.029 [-0.051 to -0.007] | -0.010 [-0.034 to 0.014] | -0.020 [-0.036 to -0.003] | -0.019 [-0.042 to 0.005]
  Week 24 (N: 22, 20, 42, 21) | -0.057 [-0.081 to -0.034] | -0.037 [-0.062 to -0.012] | -0.047 [-0.064 to -0.030] | -0.040 [-0.064 to -0.015]
  Week 50 (N: 22, 19, 41, 18) | -0.119 [-0.152 to -0.086] | -0.080 [-0.115 to -0.045] | -0.099 [-0.124 to -0.075] | -0.107 [-0.142 to -0.072]
  Week 76 (N: 22, 17, 39, 16) | -0.163 [-0.213 to -0.114] | -0.117 [-0.171 to -0.064] | -0.140 [-0.177 to -0.104] | -0.157 [-0.211 to -0.102]
  Week 104 (N: 18, 16, 34, 14) | -0.222 [-0.288 to -0.155] | -0.158 [-0.230 to -0.086] | -0.190 [-0.239 to -0.140] | -0.230 [-0.305 to -0.155]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline left hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 10; Test type: Superiority or Other; p = 0.5134, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.011, 95% CI 2-sided [-0.043 to 0.022]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.6083, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.024 to 0.041]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.9401, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.029 to 0.027]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline left hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p = 0.2950, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.051 to 0.016]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.8817, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.031 to 0.037]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.6072, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.037 to 0.022]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline left hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 50; Test type: Superiority or Other; p = 0.6259, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.060 to 0.036]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.2807, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.023 to 0.076]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.7224, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 0.008, 95% CI 2-sided [-0.035 to 0.050]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline left hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 76; Test type: Superiority or Other; p = 0.8532, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.080 to 0.067]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.3116, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.038 to 0.116]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.6246, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.049 to 0.082]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline left hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.8697, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.092 to 0.108]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p = 0.1707, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.072, 95% CI 2-sided [-0.032 to 0.176]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p = 0.3732, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.049 to 0.129]

11. Other Pre Specified Outcome: Change From Baseline in Volumetric Brain MRI Measurements in HBSI, Right
Description: Right HBSI measures the right hippocampal atrophy from registered MRI scan pairs, by subtracting the corresponding area under the intensity profile across a boundary in the repeat scans.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
mL
  Week 10 (N: 22, 20, 42, 20) | -0.027 [-0.051 to -0.004] | -0.005 [-0.030 to 0.020] | -0.016 [-0.033 to 0.001] | -0.021 [-0.046 to 0.003]
  Week 24 (N: 22, 20, 42, 21) | -0.067 [-0.091 to -0.044] | -0.027 [-0.052 to -0.002] | -0.047 [-0.064 to -0.030] | -0.059 [-0.084 to -0.035]
  Week 50 (N: 22, 19, 41, 18) | -0.133 [-0.168 to -0.098] | -0.078 [-0.116 to -0.041] | -0.106 [-0.132 to -0.080] | -0.119 [-0.157 to -0.081]
  Week 76 (N: 22, 17, 39, 16) | -0.194 [-0.252 to -0.135] | -0.136 [-0.199 to -0.072] | -0.165 [-0.208 to -0.121] | -0.177 [-0.242 to -0.113]
  Week 104 (N: 18, 16, 34, 14) | -0.247 [-0.318 to -0.175] | -0.170 [-0.247 to -0.093] | -0.208 [-0.261 to -0.156] | -0.240 [-0.320 to -0.161]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline right hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 10; Test type: Superiority or Other; p = 0.7259, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.040 to 0.028]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.3517, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.018 to 0.051]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.7311, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.024 to 0.035]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline right hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 24; Test type: Superiority or Other; p = 0.6446, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.041 to 0.026]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.0640, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.002 to 0.066]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.4057, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.017 to 0.041]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline right hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 50; Test type: Superiority or Other; p = 0.5742, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.066 to 0.037]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.1336, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.013 to 0.093]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.5734, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 0.013, 95% CI 2-sided [-0.033 to 0.058]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline right hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 76; Test type: Superiority or Other; p = 0.7067, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.016, 95% CI 2-sided [-0.104 to 0.071]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p = 0.3600, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.049 to 0.132]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p = 0.7454, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.065 to 0.090]
Statistical Analysis 13: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with baseline right hippocampal volume and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 104; Test type: Superiority or Other; p = 0.9037, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.113 to 0.100]
Statistical Analysis 14: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority or Other; p = 0.2082, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.040 to 0.181]
Statistical Analysis 15: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority or Other; p = 0.5044, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.063 to 0.127]

12. Other Pre Specified Outcome: Change From Baseline in Neuropsychological Test Battery (NTB)
Description: The NTB evaluated cognitive domains that are known to be affected early in the course of Alzheimer's disease (AD). The cognitive tests included in the NTB were: Rey Auditory Verbal Learning Test - Immediate recall, Detection, Identification, Go-No-Go Task, One Back Task, Controlled Oral Word Association Test, Category Fluency Test, and Rey Auditory Verbal Learning Test - delayed recall and recognition. For each of the eight NTB components, an individual z-score was derived based on the primary raw score of each test. Based on the individual z-scores, a composite z-score was derived using the formula: (z1-z2-z3-z4+z5+z6+z7+z8)/8. Positive change indicating an improvement from baseline.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-scores
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
z-scores
  Week 26 (N: 20, 20, 40, 19) | -0.14 [-0.28 to 0.00] | -0.07 [-0.21 to 0.08] | -0.10 [-0.20 to 0.00] | -0.11 [-0.25 to 0.04]
  Week 52 (N: 22, 19, 41, 20) | -0.08 [-0.26 to 0.09] | -0.08 [-0.27 to 0.11] | -0.08 [-0.21 to 0.05] | -0.06 [-0.25 to 0.12]
  Week 78 (N: 22, 18, 40, 18) | -0.31 [-0.52 to -0.10] | 0.01 [-0.22 to 0.23] | -0.15 [-0.31 to 0.00] | -0.27 [-0.50 to -0.04]
  Week 104 (N: 18, 18, 36, 15) | -0.42 [-0.71 to -0.14] | -0.12 [-0.42 to 0.18] | -0.27 [-0.48 to -0.06] | -0.45 [-0.76 to -0.14]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.7687, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.23 to 0.17]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.6804, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.16 to 0.24]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9452, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.17 to 0.18]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.8825, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.27 to 0.23]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.8791, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.28 to 0.24]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.8628, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.02, 95% CI 2-sided [-0.24 to 0.20]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.7843, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.35 to 0.26]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0857, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.04 to 0.60]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.3878, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.15 to 0.39]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.8918, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.39 to 0.45]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.1233, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.09 to 0.76]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.3302, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.19 to 0.55]

13. Other Pre Specified Outcome: Change From Baseline in Functional Activities Questionnaire (FAQ) Total Score
Description: FAQ is a 10-item, caregiver-based questionnaire and was administered to the study partner who was asked to rate the participant's ability to perform a variety of activities ranging from shopping, doing the laundry, simple financial transactions, comprehension of current events, some recreational or avocational activities, and reading. FAQ total score was calculated by adding the scores from each of the 10 items. A negative change indicated an improvement from baseline. FAQ Total Score is the sum of 10 items, ranging from 0 (best possible outcome) to 100 (worst possible outcome).
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 26 (N: 22, 20, 42, 19) | 3.45 [1.89 to 5.02] | 0.25 [-1.44 to 1.94] | 1.85 [0.68 to 3.03] | 1.80 [0.02 to 3.58]
  Week 52 (N: 22, 19, 41, 19) | 4.63 [2.71 to 6.55] | 0.98 [-1.10 to 3.06] | 2.81 [1.37 to 4.24] | 2.85 [0.71 to 4.99]
  Week 78 (N: 22, 18, 40, 17) | 5.36 [3.03 to 7.69] | 2.09 [-0.45 to 4.64] | 3.73 [1.99 to 5.47] | 4.89 [2.26 to 7.51]
  Week 104 (N: 18, 18, 36, 14) | 6.90 [4.25 to 9.55] | 3.11 [0.33 to 5.89] | 5.01 [3.07 to 6.94] | 4.66 [1.66 to 7.66]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.1597, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.65, 95% CI 2-sided [-0.67 to 3.97]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.2130, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-4.01 to 0.91]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9616, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-2.06 to 2.16]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.2143, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-1.06 to 4.62]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.2151, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-4.87 to 1.12]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.9704, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.05, 95% CI 2-sided [-2.61 to 2.51]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.7857, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-3.00 to 3.95]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.1323, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-6.45 to 0.87]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.4618, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-4.29 to 1.97]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.2622, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 2.24, 95% CI 2-sided [-1.74 to 6.22]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.4499, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-5.64 to 2.55]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.8454, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-3.21 to 3.91]

14. Other Pre Specified Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SOB)
Description: Clinical Dementia Rating (CDR) is a global clinical staging instrument that was administrated by a trained rater to assess a participant's level of impairment in six domains including: Memory, Orientation, Judgement and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care, based on the CDR interview. The CDR included discussions with the participant and study partner using a structured format. A CDR-SOB score was derived based on individual scores from the six domains. A negative change indicated an improvement from baseline. The total CDR-SB score is calculated as the sum of the six clinical ratings. The CDR-SOB score range for each domain is 0 to 3. The CDR-SOB total score ranges from 0 to 18, with higher scores indicating greater dementia. If any individual item is missing, then the CDR-SB is set to missing.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 26 (N: 22, 20, 42, 20) | 0.60 [0.20 to 1.00] | 0.31 [-0.11 to 0.73] | 0.46 [0.16 to 0.75] | 0.21 [-0.22 to 0.63]
  Week 52 (N: 22, 19, 41, 20) | 1.10 [0.53 to 1.66] | 0.39 [-0.21 to 0.99] | 0.74 [0.33 to 1.16] | 0.71 [0.11 to 1.31]
  Week 78 (N: 22, 18, 40, 18) | 1.71 [1.04 to 2.39] | 0.69 [-0.04 to 1.41] | 1.20 [0.70 to 1.70] | 1.25 [0.53 to 1.97]
  Week 104 (N: 17, 18, 35, 14) | 2.15 [1.32 to 2.97] | 1.23 [0.37 to 2.10] | 1.69 [1.09 to 2.29] | 1.11 [0.23 to 2.00]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.1796, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.18 to 0.96]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.7281, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.49 to 0.69]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.3347, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.26 to 0.75]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.3425, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.43 to 1.20]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.4501, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.16 to 0.52]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.9227, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = 0.04, 95% CI 2-sided [-0.68 to 0.75]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.3450, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.51 to 1.45]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.2740, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.58 to 0.45]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.9140, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.92 to 0.82]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.0923, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-0.18 to 2.24]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.8482, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.11 to 1.35]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.2840, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.49 to 1.64]

15. Other Pre Specified Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score
Description: The NPI scale assesses 12 domains (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behavior, nighttime behavior, and appetite and eating changes). The symptoms were rated on the basis of questions administered to the study partner. If a preliminary question for each domain was answered as 'Yes', each domain was rated on a 4-point frequency scale and on a 3-point severity scale. If the preliminary question was answered as 'No', the frequency, severity, and distress scales were set to zero. A negative change indicated an improvement from baseline. For each of the 12 domains, a sub-scale score is calculated as frequency*severity and ranges from 0 to 12. The NPI total score is then calculated by summing the scores of the 12 sub-scale scores. The NPI total scores ranges from 0 to 144 with higher scores indicating greater behavioral impairment. The caregiver distress score is not included in the NPI total score.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 26 (N: 22, 20, 42, 20) | 1.51 [-0.50 to 3.52] | -0.76 [-2.87 to 1.35] | 0.38 [-1.09 to 1.84] | 3.50 [1.37 to 5.64]
  Week 52 (N: 22, 19, 41, 20) | 1.97 [-0.31 to 4.25] | 2.44 [-0.00 to 4.89] | 2.21 [0.52 to 3.89] | 2.65 [0.24 to 5.06]
  Week 78 (N: 22, 18, 40, 18) | 2.01 [-0.15 to 4.18] | 1.17 [-1.19 to 3.53] | 1.59 [-0.02 to 320] | 3.34 [0.97 to 5.71]
  Week 104 (N: 18, 18, 36, 15) | 1.38 [-0.53 to 3.29] | 1.31 [-0.61 to 3.22] | 1.34 [-0.03 to 2.71] | 2.08 [-0.03 to 4.19]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.1767, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-4.90 to 0.92]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0057, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -4.26, 95% CI 2-sided [-7.23 to -1.29]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0176, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-5.69 to -0.57]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.6790, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-3.98 to 2.61]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.9028, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-3.62 to 3.20]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.7600, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.45, 95% CI 2-sided [-3.36 to 2.47]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.4089, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-4.51 to 1.86]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.1964, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-5.49 to 1.15]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.2234, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-4.58 to 1.09]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.6186, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-3.52 to 2.12]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.5853, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-3.60 to 2.06]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.5541, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-3.23 to 1.75]

16. Other Pre Specified Outcome: Change From Baseline in NPI Distress Score (NPI-D)
Description: The NPI scale assesses 12 domains (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behavior, nighttime behavior, and appetite and eating changes). The symptoms were rated on the basis of questions administered to the study partner. For each domain, the study partner also rated his/her own 'emotional or psychological' distress caused by the participant's behavior on a 6-point scale. The study partner NPI-D total score was calculated by summing the scores of the 12 sub-scale distress scores. A negative change indicated an improvement from baseline. The caregiver distress (NPI-D) total score is calculated by summing the scores of the 12 sub-scale distress scores. The NPI-D total scores ranges from 0 to 60 with higher scores indicating greater distress.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 26 (N: 22, 20, 42, 20) | 1.49 [0.11 to 2.87] | 0.42 [-1.03 to 1.86] | 0.95 [-0.05 to 1.96] | 1.57 [0.10 to 3.05]
  Week 52 (N: 22, 19, 41, 20) | 1.54 [0.20 to 2.88] | 1.24 [-0.20 to 2.68] | 1.39 [0.39 to 2.38] | 2.27 [0.84 to 3.71]
  Week 78 (N: 22, 18, 40, 18) | 1.45 [0.11 to 2.79] | 0.44 [-1.01 to 1.90] | 0.95 [-0.05 to 1.94] | 2.56 [1.08 to 4.03]
  Week 104 (N: 18, 18, 36, 15) | 1.73 [0.02 to 3.44] | 1.76 [0.03 to 3.48] | 1.74 [0.52 to 2.97] | 1.27 [-0.62 to 3.16]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9370, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-2.09 to 1.93]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.2597, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-3.19 to 0.88]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.4852, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.38 to 1.14]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.4542, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-2.69 to 1.22]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.3061, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-3.04 to 0.97]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.3082, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.88, 95% CI 2-sided [-2.61 to 0.84]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.2672, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-3.09 to 0.87]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0427, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.11, 95% CI 2-sided [-4.15 to -0.07]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0716, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-3.37 to 0.15]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.7184, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-2.09 to 3.00]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.7004, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-2.06 to 3.03]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.6723, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-1.77 to 2.71]

17. Other Pre Specified Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score
Description: The MMSE is a brief, structured examination of cognitive function consisting of the 11 item: Orientation-What, Orientation-Where, Registration-Objects, Attention and Calculation, Recall, Language-Naming, Language-Repetition, Language-Comprehension, Language-Reading, Language-Writing, and Language- Drawing. MMSE total score was the sum of the 11 item scores and it ranges from 0 to 30 with higher score indicating greater cognitive functioning. If any individual item is missing, then the MMSE total score is set to missing. A positive change indicating an improvement from baseline.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 26 (N: 22, 20, 42, 20) | -1.06 [-2.20 to 0.09] | -1.09 [-2.28 to 0.09] | -1.08 [-1.90 to -0.25] | -1.10 [-2.29 to 0.09]
  Week 52 (N: 22, 19, 41, 20) | -2.46 [-3.72 to -1.21] | -1.54 [-2.87 to -0.20] | -2.00 [-2.92 to -1.08] | -1.30 [-2.62 to -0.01]
  Week 78 (N: 22, 18, 40, 18) | -2.28 [-3.75 to -0.82] | -1.92 [-3.48 to -0.35] | -2.10 [-3.17 to -1.03] | -1.42 [-2.97 to -0.13]
  Week 104 (N: 19, 18, 37, 15) | -3.55 [-5.48 to -1.63] | -1.34 [-3.37 to 0.68] | -2.45 [-3.85 to -1.05] | -2.53 [-4.62 to -0.44]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9535, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.58 to 1.68]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9914, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-1.63 to 1.65]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9682, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.39 to 1.44]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.2008, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.96 to 0.64]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.7988, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-2.07 to 1.60]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.3764, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.70, 95% CI 2-sided [-2.27 to 0.87]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.4177, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-2.98 to 1.25]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.6494, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-2.67 to 1.68]
Statistical Analysis 9: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.4674, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-2.54 to 1.18]
Statistical Analysis 10: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.4709, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-3.85 to 1.81]
Statistical Analysis 11: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.4128, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-1.70 to 4.07]
Statistical Analysis 12: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.9478, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-2.41 to 2.58]

18. Other Pre Specified Outcome: Change From Baseline in 13-item Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) Total Score
Description: The ADAS-Cog is a global cognitive measure. For the following 13 items, the participants were rated: Word Recall, Commands, Construction Praxis, Delayed Word Recall Task, Naming Task, Ideational Praxis, Orientation, Word Recognition Task, Remembering Test Instructions, Spoken Language Ability, Word-Finding Difficulty in Spontaneous Speech, Comprehension, and Number Cancellation. The ADAS-cog is a structured scale that evaluates memory, orientation, attention, reasoning, language and constructional praxis. The total score was the sum of the scores from the 13 individual items. This study used a modified 85 point scale with a scoring range of 0 to 85 (13 items). Higher scores of the 13 individual items indicated greater cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
score
  Week 54 (N: 22, 19, 41, 29) | -5.58 [-7.55 to -3.61] | -6.69 [-8.83 to -4.55] | -6.14 [-7.61 to -4.67] | -5.05 [-7.21 to -2.90]
  Week 86 (N: 19, 18, 37, 17) | 1.80 [-0.04 to 3.65] | 0.28 [-1.65 to 2.22] | 1.04 [-0.31 to 2.39] | 1.56 [-0.43 to 3.55]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 54; Test type: Superiority or Other; p = 0.7146, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-3.40 to 2.35]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.2733, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.64, 95% CI 2-sided [-4.60 to 1.33]
Statistical Analysis 3: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.3969, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-3.62 to 1.46]
Statistical Analysis 4: Comparison: ACC 3 μg+QS-21 vs Placebo; A mixed effects model for repeated measures analysis was used, with the baseline assessment and ApoE4 status as covariates, and visit, treatment and visit by treatment interaction as fixed effects, with variance-covariance structure set to unstructured. Statistical analysis presented above for Week 86; Test type: Superiority or Other; p = 0.8566, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-2.43 to 2.92]
Statistical Analysis 5: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.3460, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-3.98 to 1.42]
Statistical Analysis 6: Comparison: Overall ACC + QS21 vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.6582, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Median Difference (Final Values) = -0.52, 95% CI 2-sided [-2.86 to 1.82]

19. Other Pre Specified Outcome: Change From Baseline in Dependence Scale (DS) Score
Description: An abbreviated administration (first 6 items) of the DS was used in this study. The DS is a brief study partner-completed measure which assesses the degree of support required by a subject with AD. Since the goal of treatment was to delay or arrest the processes leading to increased dependence, the DS represented a meaningful endpoint for clinical studies in AD. The dependence score was derived by summing the first 6 items of the DS. Item 1 and 2 ranged from 0 - 2 and item 3 - 6 ranged from 0 - 1. The total score was calculated by summing the score from each of the 6 items. So the total score could range from 0 - 8, with higher scores indicating greater dependence.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 0.1 (1.44) [0.20 to 1.00] | -0.4 (1.39) [-0.11 to 0.73] | 0.0 (1.65) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | -0.2 (1.60) [0.53 to 1.66] | 0.2 (1.96) [-0.21 to 0.99] | 0.1 (1.86) [0.11 to 1.31]
  Week 78 (22, 18, 18) | 0.2 (1.07) [1.04 to 2.39] | 0.3 (1.41) [-0.04 to 1.41] | -0.2 (1.93) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 0.9 (2.21) [1.32 to 2.97] | 0.6 (1.58) [0.37 to 2.10] | -0.1 (2.07) [0.23 to 2.00]

20. Other Pre Specified Outcome: Change From Baseline in Resource Utilization in Dementia (RUD) (Abbreviated) (RUD-Lite) - Primary Caregiver
Description: An abbreviated administration of the RUD (RUD-Lite) was used. The RUD-Lite is a comprehensive tool for addressing the magnitude and nature of study partner/caregiver effort in cases of dementia. Since a significant portion of care in Alzheimer's related-dementia was performed informally by the participant's friends or family, it was desirable to measure the extent of this care for use in economic evaluations of disease. The total time spent by the primary caregiver providing support on activities of daily living (ADL), instrumental activities of daily living (IADL) and supervising, respectively, was calculated in two components. Total number of days spent during the past month on each of ADL, IADL, and supervising; and: time per day during the past month on each of ADL, IADL and supervising. The total Primary Caregiver Time per month could range from 0 - 720. This was calculated by multiplying the number of days per month (30) by the number of hours per day (24).
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
hours
  Week 26 (N: 22, 20, 20) | 3.97 [-7.02 to 14.97] | -6.05 [-17.57 to 5.47] | 6.47 [-5.23 to 18.17]
  Week 52 (N: 22, 19, 20) | 16.76 [0.60 to 32.93] | -7.97 [-25.41 to 9.47] | 21.73 [4.66 to 38.79]
  Week 78 (N: 22, 18, 18) | 30.80 [-10.69 to 72.29] | -3.23 [-49.00 to 42.54] | 61.74 [15.98 to 107.51]
  Week 104 (N: 18, 18, 15) | 36.36 [15.37 to 57.34] | -5.88 [-27.65 to 15.88] | 20.31 [-2.29 to 42.92]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.7537, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-18.36 to 13.36]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.1266, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -12.51, 95% CI 2-sided [-28.86 to 3.65]
Statistical Analysis 3: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.6724, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -4.96, 95% CI 2-sided [-28.34 to 18.41]
Statistical Analysis 4: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.0170, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -29.70, 95% CI 2-sided [-53.89 to -5.50]
Statistical Analysis 5: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.3196, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -30.94, 95% CI 2-sided [-92.67 to 30.78]
Statistical Analysis 6: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.0490, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -64.97, 95% CI 2-sided [-129.64 to -0.31]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.2969, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 16.04, 95% CI 2-sided [-14.70 to 46.79]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.0973, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -26.20, 95% CI 2-sided [-57.42 to 5.03]

21. Other Pre Specified Outcome: Change From Baseline in RUD (Abbreviated) (RUD-Lite) - Other Caregivers
Description: An abbreviated administration of the RUD (RUD-Lite) was used. The RUD-Lite is a comprehensive tool for addressing the magnitude and nature of study partner/caregiver effort in cases of dementia. Since a significant portion of care in Alzheimer's related-dementia was performed informally by the participant's friends or family, it was desirable to measure the extent of this care for use in economic evaluations of disease. The total time spent by the other caregivers providing support on ADL, IADL and supervising, respectively, was calculated in two components. Total number of days spent during the past month on each of ADL, IADL and supervising; and: time per day during the past month on each of ADL, IADL, and supervising. The total Other Caregiver Time per month could range from 0 - 720. This was calculated by multiplying the number of days per month (30) by the number of hours per day (24).
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
hours
  Week 26 (N: 22, 20, 20) | 0.14 [-4.36 to 4.64] | 4.03 [-0.69 to 8.76] | 1.56 [-3.17 to 6.28]
  Week 52 (N: 22, 19, 20) | 0.72 [-2.66 to 4.10] | 3.03 [-0.52 to 6.59] | 0.01 [-3.54 to 3.55]
  Week 78 (N: 22, 18, 18) | 0.86 [-0.36 to 2.08] | 0.79 [-0.51 to 2.10] | 0.06 [-1.25 to 1.36]
  Week 104 (N: 18, 18, 15) | 2.13 [-9.20 to 13.47] | 1.58 [-10.12 to 13.27] | 9.64 [-2.67 to 21.96]
Statistical Analysis 1: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.6653, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-7.94 to 5.10]
Statistical Analysis 2: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.4613, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [-4.20 to 9.15]
Statistical Analysis 3: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.7710, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-4.18 to 5.61]
Statistical Analysis 4: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.2328, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 3.02, 95% CI 2-sided [-1.99 to 8.04]
Statistical Analysis 5: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.3693, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-0.97 to 2.58]
Statistical Analysis 6: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.4220, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-1.09 to 2.56]
Statistical Analysis 7: Comparison: ACC 3 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.3728, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -7.51, 95% CI 2-sided [-24.25 to 9.23]
Statistical Analysis 8: Comparison: ACC 10 μg+QS-21 vs Placebo; [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p = 0.3452, Mixed-Effects Model Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger was used to estimate the denominator degrees of freedom; Mean Difference (Final Values) = -8.07, 95% CI 2-sided [-25.05 to 8.91]

22. Other Pre Specified Outcome: Percentage of Participants With a Global CDR Score of Equal to or Greater Than 1 for the First Time
Description: CDR is a global clinical staging instrument that was administrated by a trained rater to assess a participant's level of impairment in six domains including: Memory, Orientation, Judgement and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care, based on the CDR interview. The CDR included discussions with the participant and study partner using a structured format. CDR global score was derived from the six domains according to a complex algorithm with emphasis on the Memory Domain score. Global CDR score = 0.5 with memory box score of 0.5. The total CDR-SB score is calculated as the sum of the six clinical ratings. The CDR-SOB score range for each domain is 0 to 3, with higher score indicating no significant function. If any individual item is missing, then the CDR-SB is set to missing.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
percentage of participants
  Week 26 | 86.4 | 70.0 | 78.6 | 80.0
  Week 52 | 0.0 | 15.0 | 7.1 | 10.0
  Week 78 | 13.6 | 0.0 | 7.1 | 0.0
  Week 104 | 0.0 | 10.0 | 4.8 | 0.0

23. Other Pre Specified Outcome: Geometric Mean Anti-Aβ IgG Enzyme-linked Immunosorbent Assay (ELISA) Titers
Description: Site personnel collecting the samples for anti-Aβ antibody titers were blinded to the participant treatment group assignment. The lower limit of quantification (LLOQ) determined for this assay was 100 U/mL. For any anti-Aβ IgG antibody level that was below the LLOQ (100 U/mL), the lower limit of detection (LLOD) defined as 0.5*LLOQ was imputed.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Geometric Mean (95% Confidence Interval); unit: U/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
U/ml
  Baseline (N: 21, 18, 39, 21) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 53.5 [46.5 to 61.6]
  Week 2 (N: 20, 20, 40, 21) | 61.5 [48.5 to 78.0] | 81.4 [53.3 to 124.2] | 70.7 [55.9 to 89.6] | 50.0 [50.0 to 50.0]
  Week 4 (N: 21, 17, 38, 21) | 59.0 [50.3 to 69.3] | 86.3 [53.3 to 139.8] | 70.0 [55.7 to 87.9] | 50.0 [50.0 to 50.0]
  Week 6 (N: 22, 20, 42, 21) | 1490.0 [577.0 to 3847.9] | 1485.3 [570.0 to 3870.0] | 1487.7 [780.5 to 2835.9] | 50.0 [50.0 to 50.0]
  Week 10 (N:22, 20, 42, 20) | 774.8 [355.7 to 1687.7] | 960.3 [453.5 to 2033.2] | 858.1 [510.3 to 1443.1] | 50.0 [50.0 to 50.0]
  Week 12 (N: 22, 18, 40, 20) | 566.4 [270.5 to 1186.1] | 536.0 [238.7 to 1204.0] | 552.5 [328.2 to 930.1] | 50.0 [50.0 to 50.0]
  Week 14 (N: 22, 20, 42, 20) | 5997.5 [3541.6 to 10156.5] | 2796.3 [1414.2 to 5529.1] | 4170.3 [2727.9 to 6375.2] | 50.0 [50.0 to 50.0]
  Week 20 (N: 21, 20, 41, 21) | 3320.9 [1855.9 to 5942.4] | 2172.9 [1106.7 to 4266.3] | 2700.2 [1757.7 to 4148.2] | 50.0 [50.0 to 50.0]
  Week 26 (N: 22, 19, 41, 20) | 1657.0 [967.3 to 2838.5] | 1739.1 [801.9 to 3771.7] | 1694.6 [1092.4 to 2628.8] | 60.7 [40.5 to 90.9]
  Week 28 (N: 22, 20, 42, 20) | 6482.5 [4247.1 to 9894.5] | 4668.3 [2371.1 to 9190.7] | 5544.3 [3802.5 to 8083.7] | 50.0 [50.0 to 50.0]
  Week 34 (N: 22, 20, 42, 20) | 3731.9 [2375.7 to 5862.5] | 5329.0 [2754.6 to 10309.3] | 4421.9 [3024.7 to 6464.5] | 50.0 [50.0 to 50.0]
  Week 52 (N: 20, 18, 38, 19) | 1322.6 [800.2 to 2185.9] | 1920.8 [983.0 to 3753.2] | 1578.3 [1060.8 to 2348.2] | 50.0 [50.0 to 50.0]
  Week 54 (N: 20, 19, 39, 19) | 6787.7 [4892.4 to 9417.2] | 12064.7 [6642.8 to 21912.2] | 8982.9 [6438.2 to 12533.3] | 50.0 [50.0 to 50.0]
  Week 60 (N: 21, 19, 40, 19) | 4130.7 [2948.4 to 5787.2] | 9665.3 [5448.3 to 17146.1] | 6185.7 [4410.2 to 8676.0] | 50.0 [50.0 to 50.0]
  Week 78 (N: 19, 14, 33, 14) | 2007.1 [1357.3 to 2967.9] | 2973.5 [1283.4 to 6889.1] | 2371.3 [1590.2 to 3536.0] | 50.0 [50.0 to 50.0]
  Week 80 (N: 19, 14, 33, 16) | 8006.3 [4636.8 to 13824.2] | 11086.8 [6331.5 to 19413.8] | 9192.0 [6303.8 to 13403.4] | 50.0 [50.0 to 50.0]
  Week 86 (N: 15, 17, 32, 14) | 6584.2 [4090.5 to 10598.3] | 10125.5 [6528.3 to 15704.9] | 8275.6 [6046.9 to 11325.9] | 50.0 [50.0 to 50.0]
  Week 104 (N: 11, 9, 20, 9) | 3960.8 [2704.6 to 5800.7] | 3513.9 [1395.3 to 8849.1] | 3753.1 [2481.5 to 5676.2] | 50.0 [50.0 to 50.0]

24. Other Pre Specified Outcome: Geometric Mean Anti-Aβ IgM ELISA Titers
Description: Site personnel collecting the samples for anti-Aβ antibody titers were blinded to the participant treatment group assignment. The LLOQ determined for this assay was 50 U/mL. For any anti-Aβ IgM antibody level that was below the LLOQ (50 U/mL), the LLOD defined as 0.5*LLOQ was imputed.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Geometric Mean (95% Confidence Interval); unit: U/ml
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Overall ACC + QS21 | Placebo
Number analyzed (Participants) | 22 | 20 | 42 | 21
U/ml
  Baseline (N: 21, 18, 39, 21) | 31.8 [25.0 to 40.4] | 33.9 [23.6 to 48.8] | 32.7 [26.8 to 40.1] | 31.6 [26.0 to 38.4]
  Week 2 (N: 20, 20, 40, 21) | 69.7 [37.9 to 128.1] | 121.0 [66.1 to 221.6] | 91.8 [60.4 to 139.6] | 30.2 [25.1 to 36.3]
  Week 4 (N: 21, 17, 38, 21) | 75.0 [41.5 to 135.6] | 141.3 [72.8 to 274.0] | 99.6 [64.6 to 153.5] | 31.0 [25.8 to 37.1]
  Week 6 (N: 22, 20, 42, 21) | 840.8 [387.9 to 1822.8] | 975.8 [482.0 to 1975.8] | 902.6 [545.1 to 1494.5] | 31.5 [26.0 to 38.3]
  Week 10 (N:22, 20, 42, 20) | 723.6 [318.9 to 1641.8] | 967.3 [397.4 to 2354.6] | 830.8 [465.9 to 1481.5] | 32.1 [25.8 to 39.9]
  Week 12 (N: 22, 18, 40, 19) | 604.2 [277.5 to 1315.6] | 611.5 [255.3 to 1464.6] | 607.5 [349.0 to 1057.4] | 32.6 [26.1 to 40.6]
  Week 14 (N: 22, 20, 42, 20) | 1232.4 [632.4 to 2401.8] | 1194.6 [502.6 to 2839.0] | 1214.2 [724.5 to 2035.0] | 32.6 [26.0 to 40.8]
  Week 20 (N: 21, 20, 41, 21) | 1060.2 [505.2 to 2224.8] | 1070.5 [456.7 to 2509.4] | 1065.2 [622.3 to 1823.3] | 31.6 [25.9 to 38.5]
  Week 26 (N: 22, 19, 41, 20) | 684.8 [361.8 to 1296.3] | 939.4 [414.8 to 2127.4] | 792.9 [485.9 to 1293.8] | 32.6 [26.1 to 40.9]
  Week 28 (N: 22, 20, 42, 20) | 1241.6 [685.5 to 2248.7] | 1117.1 [497.8 to 2506.7] | 1180.6 [735.7 to 1894.8] | 31.9 [25.9 to 39.2]
  Week 34 (N: 22, 20, 42, 20) | 953.6 [519.4 to 1750.8] | 1084.5 [456.8 to 2574.7] | 1013.9 [616.6 to 1667.2] | 32.0 [25.9 to 39.5]
  Week 52 (N: 20, 18, 38, 19) | 493.8 [269.2 to 905.8] | 522.9 [211.7 to 1291.4] | 507.4 [305.5 to 842.7] | 29.2 [24.3 to 35.0]
  Week 54 (N: 20, 19, 39, 19) | 776.5 [426.1 to 1415.0] | 1176.0 [495.4 to 2791.3] | 950.5 [575.9 to 1568.9] | 29.8 [24.2 to 36.6]
  Week 60 (N: 21, 19, 40, 19) | 782.2 [409.2 to 1495.2] | 1228.4 [471.9 to 3197.6] | 969.2 [561.7 to 1672.4] | 31.0 [24.9 to 38.7]
  Week 78 (N: 19, 14, 33, 14) | 635.3 [306.2 to 1318.2] | 321.4 [111.1 to 929.4] | 475.8 [263.4 to 859.5] | 28.5 [23.5 to 34.5]
  Week 80 (N: 19, 14, 33, 16) | 744.8 [376.0 to 1475.0] | 677.0 [213.5 to 2174.2] | 715.2 [397.0 to 1288.6] | 30.7 [23.9 to 39.3]
  Week 86 (N: 15, 17, 32, 14) | 768.1 [278.7 to 2117.0] | 1023.7 [361.0 to 2903.0] | 894.7 [449.0 to 1782.7] | 32.2 [23.7 to 43.7]
  Week 104 (N: 11, 9, 20, 9) | 602.7 [221.2 to 1642.1] | 287.8 [65.1 to 1271.9] | 432.2 [195.1 to 957.3] | 29.2 [20.4 to 41.9]

25. Other Pre Specified Outcome: Change From Baseline in Perceived Deficits Questionnaire (PDQ) - Subject - Attention/Concentration Domain Score
Description: The PDQ is a tool consisting of 20 questions and is designed to assess perceived cognitive deficits from the participant's perspective. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Attention/Concentration Domain Score is the sum of the raw scores on items 1, 5, 9, 13 and 17, with a range from 0 - 4 for each of the 5 items. So the Attention/Concentration Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 0.5 (3.07) [0.20 to 1.00] | 0.1 (2.95) [-0.11 to 0.73] | 0.5 (3.49) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 0.7 (2.41) [0.53 to 1.66] | -0.1 (2.91) [-0.21 to 0.99] | 0.7 (3.34) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 0.7 (3.27) [1.04 to 2.39] | -0.1 (2.83) [-0.04 to 1.41] | 1.4 (3.66) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 1.6 (3.54) [1.32 to 2.97] | 1.1 (3.14) [0.37 to 2.10] | 1.3 (3.79) [0.23 to 2.00]

26. Other Pre Specified Outcome: Change From Baseline in PDQ - Subject - Retrospective Memory Domain Score
Description: The PDQ is a tool consisting of 20 questions and is designed to assess perceived cognitive deficits from the participant's perspective. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Retrospective Memory Domain Score is the sum of the raw scores on items 2, 6, 10, 14, and 18, with a range from 0 - 4 for each of the 5 items. So the Retrospective Memory Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 0.5 (3.11) [0.20 to 1.00] | -1.2 (2.89) [-0.11 to 0.73] | 0.4 (4.21) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 0.0 (2.82) [0.53 to 1.66] | 0.2 (2.52) [-0.21 to 0.99] | 0.5 (4.12) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 1.0 (3.78) [1.04 to 2.39] | 0.1 (2.61) [-0.04 to 1.41] | 1.2 (4.14) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 1.6 (3.47) [1.32 to 2.97] | -0.3 (2.59) [0.37 to 2.10] | 1.4 (5.03) [0.23 to 2.00]

27. Other Pre Specified Outcome: Change From Baseline in PDQ - Subject - Prospective Memory Domain Score
Description: The PDQ is a tool consisting of 20 questions and is designed to assess perceived cognitive deficits from the participant's perspective. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Prospective Memory Domain Score is the sum of the raw scores on items 3, 7, 11, 15, and 19, with a range from 0 - 4 for each of the 5 items. So the Prospective Memory Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 0.1 (2.65) [0.20 to 1.00] | -0.1 (2.17) [-0.11 to 0.73] | -0.7 (3.48) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 0.4 (2.94) [0.53 to 1.66] | 0.1 (1.73) [-0.21 to 0.99] | -0.1 (2.70) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 0.3 (2.51) [1.04 to 2.39] | -0.1 (1.43) [-0.04 to 1.41] | 0.9 (2.80) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 0.5 (2.66) [1.32 to 2.97] | 0.6 (1.94) [0.37 to 2.10] | 1.3 (3.88) [0.23 to 2.00]

28. Other Pre Specified Outcome: Change From Baseline in PDQ - Subject - Planning/Organization Domain Score
Description: The PDQ is a tool consisting of 20 questions and is designed to assess perceived cognitive deficits from the participant's perspective. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Planning/Organization Domain Score is the sum of the raw scores on items 4, 8, 12, 16, and 20, with a range from 0 - 4 for each of the 5 items. So the Planning/Organization Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 0.3 (3.39) [0.20 to 1.00] | -0.4 (2.08) [-0.11 to 0.73] | -0.4 (3.05) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 0.3 (2.91) [0.53 to 1.66] | -0.1 (2.53) [-0.21 to 0.99] | 0.3 (3.26) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 1.0 (3.73) [1.04 to 2.39] | 1.2 (1.80) [-0.04 to 1.41] | 0.9 (4.34) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 1.6 (3.35) [1.32 to 2.97] | 1.0 (2.45) [0.37 to 2.10] | 1.3 (3.79) [0.23 to 2.00]

29. Other Pre Specified Outcome: Change From Baseline in PDQ - Subject - Total Score
Description: The PDQ is a tool consisting of 20 questions and is designed to assess perceived cognitive deficits from the participant's perspective. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Total Score is computed by adding raw scores for all of the items (or all 4 domain scores) together. It could range from 0 - 80, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 1.4 (10.72) | -1.6 (7.54) | -0.3 (12.95)
  Week 52 (N: 22, 19 , 20) | 1.5 (8.60) | 0.2 (7.83) | 1.5 (11.60)
  Week 78 (N: 22, 18, 18) | 3.0 (11.03) | 1.2 (6.53) | 4.4 (13.74)
  Week 104 (N: 18, 18,15) | 5.2 (10.76) | 2.4 (8.36) | 5.3 (15.63)

30. Other Pre Specified Outcome: Change From Baseline in PDQ-R - Relative - Attention/Concentration Domain Score
Description: The PDQ-R is a tool consisting of 20 questions, is designed to assess perceived cognitive deficits, and was administered to the study partner. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Attention/Concentration Domain Score is the sum of the raw scores on items 1, 5, 9, 13, and 17, with a range from 0 - 4 for each of the 5 items. So the Attention/Concentration Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 2.0 (3.37) [0.20 to 1.00] | -0.1 (3.85) [-0.11 to 0.73] | 0.9 (2.83) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 2.0 (3.43) [0.53 to 1.66] | -0.1 (3.85) [-0.21 to 0.99] | 1.8 (2.75) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 2.9 (3.38) [1.04 to 2.39] | 0.9 (3.77) [-0.04 to 1.41] | 2.0 (3.14) [0.53 to 1.97]
  Week 104 (N: 17, 18,15) | 3.9 (3.52) [1.32 to 2.97] | 1.1 (3.16) [0.37 to 2.10] | 1.1 (4.16) [0.23 to 2.00]

31. Other Pre Specified Outcome: Change From Baseline in PDQ-R - Relative - Retrospective Memory Domain Score
Description: The PDQ-R is a tool consisting of 20 questions, is designed to assess perceived cognitive deficits, and was administered to the study partner. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Retrospective Memory Domain Score is the sum of the raw scores on items 2, 6, 10, 14, and 18, with a range from 0 - 4 for each of the 5 items. So the Retrospective Memory Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 1.3 (3.49) [0.20 to 1.00] | 0.0 (2.83) [-0.11 to 0.73] | 1.8 (2.57) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 1.7 (2.95) [0.53 to 1.66] | 0.4 (2.55) [-0.21 to 0.99] | 1.4 (2.41) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 2.3 (2.55) [1.04 to 2.39] | 1.2 (2.57) [-0.04 to 1.41] | 2.2 (2.09) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 3.1 (3.03) [1.32 to 2.97] | 1.7 (2.89) [0.37 to 2.10] | 1.7 (3.99) [0.23 to 2.00]

32. Other Pre Specified Outcome: Change From Baseline in PDQ-R - Relative - Prospective Memory Domain Score
Description: The PDQ-R is a tool consisting of 20 questions, is designed to assess perceived cognitive deficits, and was administered to the study partner. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Prospective Memory Domain Score is the sum of the raw scores on items 3, 7, 11, 15, and 19, with a range from 0 - 4 for each of the 5 items. So the Prospective Memory Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 1.0 (2.13) [0.20 to 1.00] | -0.4 (2.08) [-0.11 to 0.73] | 1.1 (2.19) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 0.6 (2.22) [0.53 to 1.66] | 0.3 (2.51) [-0.21 to 0.99] | 1.0 (2.86) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 1.5 (2.37) [1.04 to 2.39] | 0.2 (2.53) [-0.04 to 1.41] | 0.8 (2.92) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 2.6 (2.48) [1.32 to 2.97] | 0.9 (2.31) [0.37 to 2.10] | 0.5 (3.76) [0.23 to 2.00]

33. Other Pre Specified Outcome: Change From Baseline in PDQ-R - Relative - Planning/Organization Domain Score
Description: The PDQ-R is a tool consisting of 20 questions, is designed to assess perceived cognitive deficits, and was administered to the study partner. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Planning/Organization Domain Score is the sum of the raw scores on items 4, 8, 12, 16, and 20, with a range from 0 - 4 for each of the 5 items. So the Planning/Organization Domain Score could range from 0 - 20, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 1.9 (3.07) [0.20 to 1.00] | -0.2 (2.76) [-0.11 to 0.73] | 1.7 (2.80) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 1.7 (3.28) [0.53 to 1.66] | 0.3 (4.27) [-0.21 to 0.99] | 1.7 (2.74) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 2.5 (.36) [1.04 to 2.39] | -0.1 (3.39) [-0.04 to 1.41] | 1.9 (2.91) [0.53 to 1.97]
  Week 104 (N: 18, 18,15) | 2.7 (3.87) [1.32 to 2.97] | 1.1 (3.90) [0.37 to 2.10] | 1.0 (3.63) [0.23 to 2.00]

34. Other Pre Specified Outcome: Change From Baseline in PDQ-R - Relative - Total Score
Description: The PDQ-R is a tool consisting of 20 questions, is designed to assess perceived cognitive deficits, and was administered to the study partner. The instrument assessed a variety of questions in the following areas: attention/concentration, retrospective memory, prospective memory, and planning/organization. The Total Score is computed by adding raw scores for all of the items (or all 4 domain scores) together. It could range from 0 - 80, with higher scores indicating greater perceived cognitive impairment.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 20 | 21
score
  Week 26 (N: 22, 20 , 20) | 6.2 (10.69) [0.20 to 1.00] | -0.6 (10.37) [-0.11 to 0.73] | 5.4 (8.03) [-0.22 to 0.63]
  Week 52 (N: 22, 19 , 20) | 6.0 (9.91) [0.53 to 1.66] | 0.9 (11.65) [-0.21 to 0.99] | 5.7 (7.89) [0.11 to 1.31]
  Week 78 (N: 22, 18, 18) | 9.2 (9.50) [1.04 to 2.39] | 2.2 (10.30) [-0.04 to 1.41] | 6.9 (8.90) [0.53 to 1.97]
  Week 104 (N: 17, 18,15) | 12.8 (10.59) [1.32 to 2.97] | 4.8 (9.98) [0.37 to 2.10] | 4.3 (13.68) [0.23 to 2.00]

35. Other Pre Specified Outcome: Alzheimer's Disease Medication Administration Concerns Questionnaire (AD MACQ)
Description: The AD MACQ was administered to the study partner to address preferences for medication administration by assessing: Question a: I would find it easy to give the study medication to the patient myself. Question b: The number of times the medication was given was convenient. Question c: I would prefer to have the study medication given at home by me instead of at the doctor's office by the doctor or nurse. Question d: I would prefer to have the study medication given at home by a nurse instead of at the doctor's office by the doctor or nurse. Question e: Overall, I am satisfied with the way the medication was given.
Time Frame: 104 weeks
Population: FAS population included all randomized participants who had at least one dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Number analyzed (Participants) | 22 | 19 | 20
percentage of participants
  Question a: Agree | 40.9 | 42.1 | 25
  Question a: Slightly Agree | 13.6 | 0 | 0
  Question a: Neither Agree Nor Disagree | 13.6 | 21.1 | 0
  Question a: Slightly Disagree | 9.1 | 0 | 10
  Question a: Disagree | 22.7 | 36.8 | 65
  Question b: Agree | 68.2 | 68.4 | 70
  Question b: Slightly Agree | 9.1 | 10.5 | 15
  Question b: Neither Agree Nor Disagree | 22.7 | 21.1 | 15
  Question b: Slightly Disagree | 0 | 0 | 0
  Question b: Disagree | 0 | 0 | 0
  Question c: Agree | 4.5 | 26.3 | 20
  Question c: Slightly Agree | 13.6 | 5.3 | 0
  Question c: Neither Agree Nor Disagree | 22.7 | 26.3 | 10
  Question c: Slightly Disagree | 4.5 | 0 | 10
  Question c: Disagree | 54.5 | 42.1 | 60
  Question d: Agree | 27.3 | 21.1 | 20
  Question d: Slightly Agree | 4.5 | 10.5 | 0
  Question d: Neither Agree Nor Disagree | 40.9 | 31.6 | 25
  Question d: Slightly Disagree | 0 | 5.3 | 15
  Question d: Disagree | 27.3 | 31.6 | 40
  Question e: Agree | 63.6 | 84.2 | 80
  Question e: Slightly Agree | 13.6 | 0 | 5
  Question e: Neither Agree Nor Disagree | 22.7 | 15.8 | 15
  Question e: Slightly Disagree | 0 | 0 | 0
  Question e: Disagree | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 throughout the study (104 weeks).
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | ACC 3 μg+QS-21 | ACC 10 μg+QS-21 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 6/20 | 6/21
Other Adverse Events (participants affected / at risk) | 20/22 | 19/20 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 μg+QS-21 (N=22) | ACC 10 μg+QS-21 (N=20) | Placebo (N=21)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 μg+QS-21 (N=22) | ACC 10 μg+QS-21 (N=20) | Placebo (N=21)
Injection site reaction (General disorders) | 15 | 16 | 5
Fatigue (General disorders) | 2 | 2 | 1
Asthenia (General disorders) | 1 | 1 | 1
Injection site haemorrhage (General disorders) | 3 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 2
Injection site pruritus (General disorders) | 1 | 1 | 0
Irritability (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 3
Nasopharyngitis (Infections and infestations) | 4 | 3 | 2
Bronchitis (Infections and infestations) | 1 | 3 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 1
Influenza (Infections and infestations) | 1 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 4 | 3
Dizziness (Nervous system disorders) | 3 | 3 | 2
Cerebral microhaemorrhage (Nervous system disorders) | 1 | 1 | 1
Dementia Alzheimers type (Nervous system disorders) | 2 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Nerve compression (Nervous system disorders) | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 3
Grief reaction (Psychiatric disorders) | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 1
Eye inflammation (Eye disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 2 | 0
Colon operation (Surgical and medical procedures) | 0 | 1 | 0
Dental implantation (Surgical and medical procedures) | 0 | 1 | 0
Aortic valve calcification (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
In 2013 Pfizer and Janssen Alzheimer Immunotherapy Alliance made the decision that ACC-001 would not be further developed in mild to moderate AD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.